CLINICAL TRIAL: NCT04905277
Title: Beta1-Selective Blockade for Prevention of Postmenopausal Bone Loss: A Phase 2, Multi-Center, Double-Blinded, Randomized Placebo-Controlled Trial
Brief Title: Atenolol for the Prevention of Osteoporosis (APO)
Acronym: APO
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sundeep Khosla, M.D. (Other)
Collaborators: Columbia University (Other); MaineHealth (Other); University of California, San Francisco (Other)
Responsible Party: Sponsor-Investigator, Sundeep Khosla, M.D., Dr. Francis Chucker and Nathan Landow Research Professor Distinguished Mayo Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18-005725
Record Dates: First submitted 2021-05-24; First posted 2021-05-27 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Healthy
MeSH Terms: interventions — Atenolol

STUDY DESIGN:
Intervention Model Description: Atenolol vs. Placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Atenolol (Experimental): Study subjects will take Atenolol 50 mg daily over 2 years
  Interventions: Drug: Atenolol 50 MG
- Placebo (Placebo Comparator): Study subjects will take a placebo daily over 2 years
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atenolol 50 MG — 50 mg Atenolol daily
  Other Names: Atenolol
  Arms: Atenolol
Drug: Placebo — one placebo daily
  Arms: Placebo

SUMMARY:
Evaluate whether treatment with a widely used beta blocker, atenolol, will prevent bone loss at the lower back and hip in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide informed consent
* Postmenopausal women (FSH ≥ 16 IU/L) (no menses for at least one year)
* Aged 50-75 years

Exclusion Criteria:

* Clinical diagnosis of diabetes mellitus requiring insulin
* Clinically significant abnormality in any of the additional screening laboratory studies
* A1c- ≥8
* Calcium - > upper limit lab value per site
* AST- 2x upper normal limit
* FSH- < 16IU/L
* eGFR- < 45 mL/min/1.73m2 based on creatinine
* CBC- Per PI interpretation of each patient
* Presence of (documented clinical diagnosis of any of the following):

  * Significant liver or renal disease
  * Malignancy (current diagnosis including myeloma or melanoma)
  * Radiation (the site PI will determine eligibility on a case-by-case basis)
  * Malabsorption (current clinical diagnosis or actively receiving treatment)
  * Hypoparathyroidism (current clinical diagnosis or actively receiving treatment)
  * Hyperparathyroidism (current clinical diagnosis or actively receiving treatment)
  * Acromegaly
  * Cushing syndrome
  * Hypopituitarism
  * Severe chronic obstructive pulmonary disease
  * Pheochromocytoma (current clinical diagnosis or actively receiving treatment)
  * History of cardiac failure
  * Ejection Fraction <35% (based on most recent EF within the last 12 months, if available)
  * PR interval > 200 msec on screening ECG or known heart block
  * History of bronchospastic disease with treatment (asthma, bronchitis)
  * Gastric Bypass
  * Parkinson's
  * Rheumatoid Arthritis
  * Psoriatic Arthritis
  * Connective Tissue disease
* Undergoing treatment with any medications that affect bone turnover, including the following:

  * adrenocorticosteroids (oral for > 3 months within the past year or year-round use of inhaled corticosteroid use)
  * anticonvulsant therapy for seizures (carbamazepine, phenobarbital, or phenytoin within the previous year) pharmacological doses of: thyroid hormone (causing decline of thyroid stimulating hormone below normal, i.e. < 0.3 miU/L) bisphosphonates (within the past 3 yrs; if taken orally >1 month in past 3 years) denosumab, romosozumab, estrogen therapy (does not include creams or suppositories) or treatment with a selective estrogen receptor modulator, or teriparatide/abaloparatide (> 1 month within the past year); aromatase inhibitors (>1 month within the past year)
  * Current use of digitalis glycosides
  * Thiazides (< 6 months of use prior to screening)
  * Current or within the past 3 months use of beta blockers
* Any recent fracture within the past 6 months prior to screening (other than fingers, toes and facial fractures, which are all acceptable)
* Bilateral hip replacements or metal in both hips
* Patients with serum 25-hydroxyvitamin D levels of < 20 ng/ml, in order to ensure vitamin D sufficiency
* Resting systolic blood pressure < 115 mm Hg, heart rate < 55 bpm (average of 3 readings after a 5-minute rest and one minute between readings with an automatic cuff)

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome: Percent change in total hip bone mineral density (BMD) | Baseline, 24 months
  Percent change in total hip bone mineral density (BMD) by DXA

SECONDARY OUTCOMES:
Secondary Outcomes: Percent changes in lumbar spine and femur neck BMD | Baseline, 24 months
  Percent changes in lumbar spine and femur neck BMD
Additional secondary outcomes | Baseline, intermediate timepoints, 24 months
  Percent changes in radius and ultra-distal radius BMD using DXA and in bone turnover markers (CTx, PINP).

CONTACTS AND LOCATIONS:
Overall Officials: Sundeep Khosla, MD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - MaineHealth, Scarborough, Maine
  - Mayo Clinic, Rochester, Minnesota
  - Columbia University Irving Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-11-17): https://cdn.clinicaltrials.gov/large-docs/77/NCT04905277/ICF_000.pdf